CLINICAL TRIAL: NCT00776412
Title: Biomarkers of Inflammation, Coagulation, and Endothelial Function in HIV-Infected Adults
Brief Title: Blood Markers of Inflammation, Blood Clotting and Blood Vessel Function in HIV-infected Adults
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 090013; 09-I-0013
Record Dates: First submitted 2008-10-18; First posted 2008-10-21 (Estimated); Last update posted 2025-10-02 (Actual); Status verified 2025-07-02

CONDITIONS: Inflammation; Pathologic Processes
Keywords: Immunologic Non-Responder; Cardiovascular Disease; Antiretroviral; Mortality; Natural History; HIV Positive; HIV Negative; Healthy Volunteer; HV
MeSH Terms: conditions — Inflammation; Pathologic Processes; Cardiovascular Diseases; HIV Seropositivity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- HIV negative: Healthy Volunteer cohort
- HIV positive INR: HIV positive INR cohort
- HIV positive Standard: HIV positive Standard cohort

SUMMARY:
This study will collect information about markers of inflammation, blood clotting and blood vessel function in HIV-infected adults and healthy volunteers. Biomarkers are biological indicators that have been associated with disease. Certain markers of inflammation, blood clotting, and blood vessel function have been associated with risk of cardiovascular disease, stroke and death. One marker, called D-dimer, is a breakdown product of blood clots that has been associated with serious medical conditions, including deep vein thrombosis (formation of a blood clot in a vein deep in the body) and pulmonary embolism (blockage in the pulmonary artery that occurs when a blood clot from a vein breaks away, travels to the pulmonary artery and lodges there). High D-dimer levels have also been associated with cardiovascular disease and stroke risk. In a recent study of HIV-infected patients, higher D-dimer levels were strongly correlated with risk of death from any cause. The significance of changes in D-dimer and other biomarkers in HIV-infected adults is not well understood. This study will further explore D-dimer and other biomarkers to try to better understand the relationships between them and HIV infection.

Healthy volunteers and HIV-infected adults 18 years of age or older may be eligible for this study. Two visits are involved, as follows:

Visit 1 (screening visit to determine eligibility)

* Medical history and physical examination.
* Blood tests for HIV infection, blood counts, liver and kidney function.
* Pregnancy test for women who can become pregnant.

Visit 2

* Blood tests for hepatitis B and C
* Blood tests for markers of inflammation and blood clotting.
* Blood test for genetic changes that influence blood clotting.

In some cases, visits 1 and 2 may be combined.

Optional additional visits (up to 8 visits over 3 years)

* Additional blood draws for investigation of specific clinical or laboratory findings may be requested.

DETAILED DESCRIPTION:
D-dimer, a fibrin degradation product generated as a result of plasmin mediated clot dissolution processes, is an indicator of recent clot formation and subsequent fibrinolysis. Analysis of D-dimer concentration is employed in the diagnosis of deep vein thrombosis, pulmonary embolism, and disseminated intravascular coagulation. More recently, D-dimer levels have been correlated with atherosclerotic cardiovascular disease. In a recent case-control study of biomarkers for cardiovascular disease in human immunodeficiency virus (HIV)-infected adults, baseline D-dimer levels strongly correlated with all-cause mortality. Notably, the association between baseline D-dimer levels and death due to cardiovascular disease was less significant.

At present, the pathophysiology underlying the association of elevated D-dimer concentrations with mortality in HIV is not understood. This study seeks to identify possible mechanisms underlying D-dimer elevations in HIV-infected adults by investigating a number of pathways that may be associated with the elevations using biomarkers of inflammation, hemostasis, thrombosis, platelet function, lipid metabolism, and additional indicators of endothelial function. Further elucidation of plausible pathways contributing to D-dimer elevation could, ultimately, lead to trials of risk-reducing interventions for patients with an elevated D-dimer level.

This study, an exploratory, cross-sectional study of up to 350 subjects, seeks to prospectively collect data on D-dimer and related biomarkers in HIV-infected adults. Initially, the study will recruit HIV-infected adults with HIV viremia who are not taking antiretroviral therapy (ART) and compare their clinical histories and biomarker findings with those from (1) a group of HIV-infected adults with controlled HIV viremia who are receiving ART, and with those from (2) a control group of HIV-negative healthy subjects. Additionally, to study the impact of persistent immune activation and inflammation on immune responses to ART, a cohort of HIV-infected adults with poor CD4+ cell recovery despite effective ART, and to better understand the mechanisms that contribute to impaired immunologic recovery, a cohort of HIV-infected adults with poor CD4+ cell recovery despite effective ART will be enrolled (immunologic non-responder cohort) and for comparison, a control group with similar nadir CD4 counts but with good CD4+ cell recovery on ART.

The study requires 2 visits for screening, history and physical examination, and phlebotomy. A wide array of research assays investigating different aspects of inflammation, coagulation, and endothelial function will be completed. Samples will be stored for future investigation.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Age greater than or equal to 18 years
* Ability to understand and provide informed consent
* Adequate venous access
* Adequate blood counts (hemoglobin greater than or equal to 9.0 g/dL, platelets greater than or equal to 50,000 cells/mm(3))
* Willing and able to comply with study requirements and procedures including storage of blood samples for use in future studies of HIV, AIDS, immune function, inflammation, coagulation, and atherosclerosis
* Negative serum pregnancy test for females of child-bearing potential (female subjects who have medical documentation of hysterectomy and/or bilateral oophorectomy do not need to undergo pregnancy testing)

For HIV-negative subjects:

- No known history of HIV infection. At enrollment, HIV antibody testing will be performed to confirm negative HIV-1 antibody status.

For HIV-positive subjects:

* Established HIV diagnosis (previous documentation of HIV-1 infection in the subject s medical record; for subjects without such confirmation, positive ELISA testing confirmed by Western Blot or other confirmatory test, or plasma HIV viral load greater than 10,000 copies/mL)
* Must be under the care of a physician for HIV and general medical issues.

For HIV-positive subjects enrolling in the immunologic non-responder cohort:

* CD4 count less than 300 cells/mm(3) after two years of effective combination ART with documentation of viral suppression
* HIV viral load less than 50 copies/mL at screening, with no viral load greater than 1,000 copies/ml during the period of viral suppression.
* Not currently receiving any medication known to be associated with a low CD4 count
* No concurrent illness known to cause a low CD4 count
* Controls for this cohort will have a historical nadir CD4 count less than 300 cells/mm3, with current CD4 count greater than 300 cells/mm3 after three years of effective combination ART with documentation of viral suppression.

EXCLUSION CRITERIA:

* Pregnant or breast-feeding
* Known bleeding or clotting disorder
* Current use of prescription anticoagulant including warfarin, low molecular weight heparin, clopidogrel or platelet aggregation inhibitor
* Concurrent malignancy requiring cytotoxic chemotherapy or radiation therapy
* Substance abuse or severe psychiatric disorder that would interfere with adherence to protocol requirements
* Any serious medical condition for which the principal investigator feels participation may be contraindicated

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV positive patients and HIV negative healthy controls will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 310 (Actual)
Dates: Start 2008-11-20 (Actual)

PRIMARY OUTCOMES:
Obtain blood samples for further investigation into the correlation between markers of coagulation, including D-dimer, and markers of platelet function, inflammation, endothelial cell function, and clinical parameters in HIV-infected adults. | Cross-sectional and longitudinal
  The findings of this exploratory study will be used to generate hypotheses for future research studies.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph A Kovacs, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kuller LH, Tracy R, Belloso W, De Wit S, Drummond F, Lane HC, Ledergerber B, Lundgren J, Neuhaus J, Nixon D, Paton NI, Neaton JD; INSIGHT SMART Study Group. Inflammatory and coagulation biomarkers and mortality in patients with HIV infection. PLoS Med. 2008 Oct 21;5(10):e203. doi: 10.1371/journal.pmed.0050203. PMID 18942885
- [Background] Borges AH, O'Connor JL, Phillips AN, Baker JV, Vjecha MJ, Losso MH, Klinker H, Lopardo G, Williams I, Lundgren JD; INSIGHT SMART Study Group; ESPRIT Study Group; SILCAAT Scientific Committee. Factors associated with D-dimer levels in HIV-infected individuals. PLoS One. 2014 Mar 13;9(3):e90978. doi: 10.1371/journal.pone.0090978. eCollection 2014. PMID 24626096
- [Background] Tenorio AR, Zheng Y, Bosch RJ, Krishnan S, Rodriguez B, Hunt PW, Plants J, Seth A, Wilson CC, Deeks SG, Lederman MM, Landay AL. Soluble markers of inflammation and coagulation but not T-cell activation predict non-AIDS-defining morbid events during suppressive antiretroviral treatment. J Infect Dis. 2014 Oct 15;210(8):1248-59. doi: 10.1093/infdis/jiu254. Epub 2014 May 1. PMID 24795473
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2009-I-0013.html